CLINICAL TRIAL: NCT01368419
Title: Phase II Study of Continuous Endostar Infusion Combined With Radiotherapy in Esophageal Cancer Patients
Brief Title: Continuous Endostar Infusion Combined With Radiotherapy in Esophageal Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Collaborators: The First People's Hospital of Lianyungang (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Endu-201105
Record Dates: First submitted 2011-06-01; First posted 2011-06-08 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: Esophageal Cancer
Keywords: Endostar; Radiotherapy; Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — endostar protein; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: Endostar; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Endostar — 75mg Endostar in 235mL normal saline, 24h continuous infusion, 6 weeks
Radiation: Radiotherapy — 6～15MV X-ray, 2Gy/time，5times/week，6 weeks

SUMMARY:
This study is to explore the clinical efficacy of continuous Endostar infusion combined with radiotherapy in esophageal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of previously untreated stage I-III esophageal cancer
* Measurable disease according to RECIST criteria
* ECOG Performance Status 0-1
* The length of esophageal carcinoma ≤ 10 cm
* Hematologic function: WBC ≥ 4.0×109/L, PLT ≥ 80×109/L, Hb ≥ 90g/L
* Renal function: Cr ≤ 2.0×UNL
* Hepatic function: BIL ≤ 2.0×UNL, ALT/AST ≤ 5.0×UNL

Exclusion Criteria:

* Pregnant or lactating women
* Evidence of bleeding diathesis, serious infection
* Serious cardiovascular disease (congestive heart failure, uncontrollable arrhythmia, unstable angina, myocardial infarction, serious heart valve disease, resistant hypertension)
* Uncontrollable mental and nervous disorders

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-05; Primary Completion 2013-05 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 1 month after treatment

SECONDARY OUTCOMES:
Overall Survival (OS) | 2 years
Time to Progression (TTP) | every three months until disease progression
Clinical Benefit Rate (CBR) | 1 month after treatment
Serum VEGF Levels | at baseline and 6 weeks
Incidence of Adverse Events | up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Xiaodong Jiang, MD, Principal Investigator — The First People's Hospital of Lianyungang
Locations (1):
- The First People's Hospital of Lianyungang, Lianyungang, Jiangsu, China